CLINICAL TRIAL: NCT03554096
Title: Brain Penetrance of 2-Hydroxybenzylamine in Humans
Brief Title: Brain Penetrance of 2-HOBA in Humans
Acronym: 2-HOBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Vanderbilt University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John Rathmacher, PhD, Director of Clinical Research, Metabolic Technologies Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MTI2018-CS03; R44AG055184 (NIH)
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Healthy Adults
Keywords: Multiple Dosage
MeSH Terms: interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Masking Description: The dietary supplement will be delivered to the Clinical Research Center by the Investigational Pharmacy at Vanderbilt University Medical Center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-HOBA (Experimental): 2-Hydroxybenzylamine acetate: 550mg dose
  Interventions: Dietary Supplement: 2-HOBA

INTERVENTIONS:
Dietary Supplement: 2-HOBA — 2-HOBA is a compound found in buckwheat and is given as 2-HOBA acetate
  Other Names: 2-Hydroxybenzylamine

SUMMARY:
The purpose of this study is to confirm that 2-HOBA crosses the blood brain barrier and to compare blood and cerebrospinal fluid levels of 2-HOBA after a single oral dose.

DETAILED DESCRIPTION:
Consenting volunteers between 40 and 70 years old with no morbidity, including males, and females who are not pregnant will be recruited for the study. Three volunteers will be enrolled with a reasonable sampling of ethnicities from the Nashville area, and an effort will be made to recruit males and females. The study will be conducted by the Vanderbilt Clinical Research Center (CRC).

Briefly, the three volunteers will be studied at a single dose level. Baseline assessments will be performed, and then each volunteer will be given a single oral dose (550 mg) of 2-HOBA. Ninety minutes after the dose, a lumbar puncture will be performed to obtain cerebrospinal fluid and a blood sample will be collected. 2-HOBA levels will be measured in cerebrospinal fluid and blood samples from this timepoint to assess the ability or orally ingested 2-HOBA to cross the blood brain barrier.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between 40 and 70 years old;
* Men and women who are not pregnant at the time of study; and
* Not taking any medication 24 hours prior to and during the study.

Exclusion Criteria:

* Inability to give informed consent;
* Current use of anticoagulant medications, such as warfarin (Coumadin), dabigatran (Pradaxa), or rivaroxaban (Xarelto), due to high risk of bleeding complications. Volunteers taking aspirin or clopidogrel (Plavix), will not be excluded, but will be asked to get clearance from their prescribing physician before stopping the drug 24 hours prior to the procedure;
* Need to discontinue any drug that is administered as standard of care treatment;
* Unwillingness or inability to use approved birth-control methods (pre-menopausal women); and
* History of lumbar surgery, fibromyalgia, current lower back pain, or scoliosis.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Brain Penetrance | 90 minutes
  Ratio of 2-HOBA concentration in the cerebrospinal fluid to plasma 2-HOBA concentration after oral administration (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pitchford LM, Driver PM, Fuller JC Jr, Akers WS, Abumrad NN, Amarnath V, Milne GL, Chen SC, Ye F, Roberts LJ 2nd, Shoemaker MB, Oates JA, Rathmacher JA, Boutaud O. Safety, tolerability, and pharmacokinetics of repeated oral doses of 2-hydroxybenzylamine acetate in healthy volunteers: a double-blind, randomized, placebo-controlled clinical trial. BMC Pharmacol Toxicol. 2020 Jan 6;21(1):3. doi: 10.1186/s40360-020-0382-y. PMID 31907026